CLINICAL TRIAL: NCT05534893
Title: Immune Benefits of Blueberry Consumption in Overweight Older Men and Postmenopausal Women: A Randomized Trial
Brief Title: Effect of Blueberries on Immunity
Acronym: Blueberry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5220098
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Immune Response; Inflammation
Keywords: Blueberries; Immunity; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This will be a parallel, free-living, randomized controlled trial, where 52 overweight men and postmenopausal women will be randomized to receive either the freeze dried blueberries or a placebo powder
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, participant, care provider, outcomes assessor will not be aware of which participant is in which arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry powder group (Experimental): Participants in the blueberry powder group will receive freeze dried blueberries in form of a powder
  Interventions: Dietary Supplement: Blueberry powder group; Dietary Supplement: Placebo powder group
- Placebo powder group (Placebo Comparator): Participants in the placebo group will receive an isocaloric placebo powder.
  Interventions: Dietary Supplement: Blueberry powder group; Dietary Supplement: Placebo powder group

INTERVENTIONS:
Dietary Supplement: Blueberry powder group — Participants in the blueberry powder group will receive freeze dried blueberries in form of a powder
Dietary Supplement: Placebo powder group — Participants in the placebo powder group will receive an isocaloric placebo powder

SUMMARY:
This research study will test the effects of Blueberries on immune functions in overweight older men and postmenopausal women

DETAILED DESCRIPTION:
This study will examine the effects of Blueberries on clinically relevant markers of immune function. Eligible and selected participants will be randomized to one of two groups at the baseline clinic visit. The Blueberry group participants will consume blueberries (2 packets of blueberry freeze-dried powder equivalent to 2 cups of fresh blueberries) added to the habitual diet and the Control group participants will abstain from blueberries (with instructions to limit the consumption of other berries and polyphenol rich foods) but otherwise continue their habitual diet. During the study, clinic visits will occur at 4-week intervals (baseline, weeks 4, 8 and 12) for a total of 4 visits at the Loma Linda University Nutrition Research Center. Blood samples taken at baseline and at week 12 will be assayed for changes in immune function and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Older men and post-menopausal women aged 50-70 year
2. Have BMI of 25-32
3. Able to commute to Loma Linda University
4. Consuming a typical American Diet low in polyphenols

Exclusion Criteria:

1. Intolerance or allergy to Blueberries
2. Regular intake of Blueberries and other berried (>2 ounces/week)
3. Immune system insufficiency or disease
4. Using immune boosting supplements
5. Exposure to antibiotics and corticoids immediately prior to study
6. Uncontrolled chronic diseases and relevant psychiatric illness, including major depression
7. Flu vaccination and or Covid Vaccination less than 3 months ago from the start of the study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
changes in lymphocyte populations | baseline to 12 weeks
  Immunophenotyping will be performed by flow cytometry to measure the number of T helper, T cytotoxic, Naïve and memory cells and B cells
changes in cytokine production | baseline to 12 weeks
  PBMC cells will be separated from blood, activated and cultured using phytohemagglutinin (PHA). Inflammatory cytokine production will be measured in the resulting supernatant using ELISA
changes in natural killer (NK) cell activity | baseline to 12 weeks
  The NK degranulation assay will be performed on blood samples. The test will be conducted using a modified flow cytometry method that measures the expression of CD107a
changes in serum inflammatory cytokine concentration | baseline to 12 weeks
  Changes in the concentrations of the inflammatory cytokines will be performed on serum using enzyme-linked immunoassay (ELISA)
changes in complete blood count (CBC) | baseline to 12 weeks
  changes in the complete blood count will be performed on whole blood with the use of an automated hematology analyzer at a certified clinical facility

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPH, Principal Investigator — Loma Linda University; Sujatha Rajaram, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No